CLINICAL TRIAL: NCT02587663
Title: Sonography Compared With MRI in Pre-Operative Evaluation of Patients With Breast Cancer to Determine Extent of Breast Disease
Brief Title: Extent of Breast Cancer and the Role of Pre-Operative Sonography and MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1B-05-5; NCI-2011-01365 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1B-05-5 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2015-09-13; First posted 2015-10-27 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Ductal Breast Carcinoma In Situ; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms | interventions — High-Energy Shock Waves; Gadolinium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (standard of care) (Active Comparator): Patients undergo standard of care diagnostic imaging comprising bilateral mammography and targeted breast ultrasound.
  Interventions: Procedure: Mammography; Procedure: Therapeutic Conventional Surgery; Procedure: Ultrasonography
- Group 2 (bilateral whole-breast ultrasound) (Experimental): Patients undergo standard of care diagnostic imaging as in Group 1. Patients also undergo bilateral whole-breast ultrasound.
  Interventions: Procedure: Mammography; Procedure: Therapeutic Conventional Surgery; Procedure: Ultrasonography
- Group 3 (bilateral breast contrast-enhanced MRI) (Experimental): Patients undergo standard of care diagnostic imaging as in Group 1. Patients also undergo bilateral breast contrast-enhanced MRI.
  Interventions: Procedure: Contrast-enhanced Magnetic Resonance Imaging; Procedure: Mammography; Procedure: Therapeutic Conventional Surgery; Procedure: Ultrasonography; Other: Gadolinium

INTERVENTIONS:
Procedure: Contrast-enhanced Magnetic Resonance Imaging — Undergo bilateral breast contrast enhanced MRI
  Other Names: CONTRAST ENHANCED MRI; Contrast-enhanced MRI
  Arms: Group 3 (bilateral breast contrast-enhanced MRI)
Procedure: Mammography — Undergo bilateral mammography
Procedure: Therapeutic Conventional Surgery — Undergo breast conserving surgery
Procedure: Ultrasonography — Undergo bilateral whole-breast ultrasound
  Other Names: ULTRASOUND; Ultrasound Imaging; Ultrasound Test; Ultrasound, Medical; US
  Arms: Group 2 (bilateral whole-breast ultrasound)
Procedure: Ultrasonography — Undergo targeted breast ultrasound
  Other Names: ULTRASOUND; Ultrasound Imaging; Ultrasound Test; Ultrasound, Medical; US
Other: Gadolinium — Contrast agent used in MRI
  Other Names: GBCA
  Arms: Group 3 (bilateral breast contrast-enhanced MRI)

SUMMARY:
This clinical trial studies mammography and targeted ultrasound with or without whole-breast ultrasound or contrast-enhanced magnetic resonance imaging (MRI) in finding out the extent of disease before surgery in patients with newly diagnosed breast cancer. New diagnostic imaging procedures, such as whole-breast ultrasound or contrast-enhanced MRI, may help find out how far breast cancer has spread. It is not yet known whether mammography and targeted ultrasound are more effective with or without whole-breast ultrasound or contrast-enhanced MRI in finding out how far breast cancer has spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine how surgical treatment is influenced by the three imaging arms.

II. To compare three imaging arms in terms of accurately measuring the size of the index lesion and the number and location of tumor foci (using surgical pathology as gold standard).

SECONDARY OBJECTIVES:

I. In women with dense breasts: To retrospectively compare the accuracy of three imaging arms in measuring the size of the index lesion and the number and location of tumor foci (using surgical pathology as the gold standard).

II. To report the incidence of synchronous contralateral breast cancers detected by the three imaging arms.

OUTLINE: Patients are assigned to 1 of 3 treatment groups.

GROUP 1: Patients undergo standard of care diagnostic imaging comprising bilateral mammography and targeted breast ultrasound.

GROUP 2: Patients undergo standard of care diagnostic imaging as in Group 1. Patients also undergo bilateral whole-breast ultrasound.

GROUP 3: Patients undergo standard of care diagnostic imaging as in Group 1. Patients also undergo bilateral breast contrast-enhanced MRI.

All patients undergo standard of care breast conserving surgery, or mastectomy if the tests indicate a change in the surgical plan.

ELIGIBILITY:
Inclusion Criteria:

* Competent to provide informed consent
* Pathologically proven invasive breast cancer or ductal carcinoma in situ (DCIS) originally identified clinically or mammographically and diagnosed by percutaneous core biopsy
* Eligible for breast conserving surgery followed by radiation therapy

Exclusion Criteria:

* Women with surgical excisional biopsy that diagnosed the breast cancer
* Women with clinical or mammographic findings where breast conserving surgery is not an option
* Women that clinically or mammographically have breast cancers that are fixed to skin
* Women receiving neoadjuvant chemotherapy prior to surgery
* Women having contraindications to contrast-enhanced (CE)-MRI examination (e.g., claustrophobia and allergy to gadolinium)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2005-11-20 (Actual); Primary Completion 2011-11-20 (Actual); Study Completion 2012-11-20 (Actual)

PRIMARY OUTCOMES:
Difference between the longest diameter of the index lesion as determined by imaging versus as determined by the pathologist | Up to 4 weeks
  Every attempt will be made to identify a transformation for the difference in the lengths of the largest diameters. If none are found, then the data will be summarized with histograms, medians, quartiles, and ranges. If a transformation is found, means, standard deviations, and 95% confidence intervals will be reported instead of the median and quartiles. Differences between three imaging methods will be compared using a paired t-test (or paired rank sum test).

SECONDARY OUTCOMES:
Number of patients identified with invasive breast cancer in women who have dense or no dense breasts as determined by the 3 imaging arms | Up to 4 weeks
  The analyses above will be rerun, stratifying by breast density: the differences in the modalities will be estimated for women with dense breasts and without, and the differences between the two groups of women will also be estimated. Dense will be defined as dense parenchyma involving more than 50% of breast volume.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Hovanessian-Larsen, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States